CLINICAL TRIAL: NCT00603785
Title: Effects of Anti-IgE Antibody Omalizumab (Xolair) on Patients With Chronic Sinusitis and a Positive Allergen Test
Brief Title: Effects of Anti-IgE Antibody Omalizumab on Patients With Chronic Sinusitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient funds available
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07030836; BB-IND# 12452
Record Dates: First submitted 2008-01-11; First posted 2008-01-29 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Chronic Sinusitis
Keywords: Chronic sinusitis; Xolair; Nasal Discharge; Nasal Obstruction; Facial Pain; Hyposmia
MeSH Terms: conditions — Rhinitis; Nasal Obstruction; Facial Pain; Anosmia | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Subjects to receive placebo treatment for 6 months
  Interventions: Drug: Placebo
- B (Experimental): Subjects to receive Xolair treatment for 6 months
  Interventions: Drug: Xolair

INTERVENTIONS:
Drug: Placebo — Subjects with chronic sinusitis and evidence of atopy and an elevated total IgE (>30 and <700 IU/ml) will be randomized to receive placebo treatment for 6 months.
  Arms: A
Drug: Xolair — Subjects with chronic sinusitis and evidence of atopy and an elevated total IgE (>30 and <700 IU/ml) will be randomized to receive Xolair treatment for 6 months.
  Arms: B

SUMMARY:
We propose to study the effects of Xolair on patients with chronic sinusitis with or without nasal polyps. Because of the similarities between the inflammatory processes found in asthmas and rhinitis to those found in chronic sinusitis, we hypothesize that sinusitis should respond to Xolair, just as asthma.

DETAILED DESCRIPTION:
We propose to study the effects of Xolair on patients with chronic sinusitis with or without nasal polyps. Since Xolair has been shown to be effective in asthmatic subjects with evidence of atopy and elevated IgE, we will limit our study to patients with chronic sinusitis and these parameters. The primary objective is to determine if Xolair decreases mucosal thickness on CT scan after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 75 years of age
* Chronic sinusitis as defined by symptoms for greater than 12 weeks despite treatment.
* Paranasal sinus CT scan showing evidence of chronic sinusitis.
* Positive skin or RAST test to an inhalant allergen.
* Serum total IgE between 30 and 700 International Units/ml.
* Body weight less than 150kg.
* Impaired quality of life as measured by the Rhinosinusitis Disability Index (RSDI).

Exclusion Criteria:

* Women of childbearing potential not using the contraception method(s) (Birth control pills, depo Provera, double barrier) as well as women who are breastfeeding.
* Known sensitivity to Xolair
* Patients with severe medical conditions that in the view of the investigator prohibits participation in the study (heart, lung, kidney, neurological, oncologic or liver disease).
* Use of any other investigational agent in the last 30 days.
* No measurable disability on the RSDI.
* Immunocompromised patients or patients with ciliary disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Estimated); Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Subjects will have QOL measures (RSDI, SNOT 20, SF-36), NPIF, and nasal lavage repeated. Exacerbations of sinusitis requiring additional treatments will be recorded. Paranasal sinus CT scans will be obtained at the screening and final visits | At entry and every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Goldberg, MD, Principal Investigator — University of California, San Francisco